CLINICAL TRIAL: NCT07036510
Title: Early Feasibility, Open-Label, Dose-Escalating, Non-Randomized Study to Evaluate the Safety of a New Timolol Sustained-Release Intraocular Implant (TimoD) in Participants With Open-Angle Glaucoma (OAG) or Ocular Hypertension (OHT) Undergoing Cataract Surgery
Brief Title: Safety of TimoD Sustained-Release Implant in Participants With Glaucoma or Ocular Hypertension Undergoing Cataract Surgery
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EyeD Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: EyeD-010-006; U1111-1317-3395 (Other: WHO)
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular hypertension; OHT; Cataract; Timolol; Lens diseases
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Cataract; Lens Diseases | interventions — Drugs, Investigational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TimoD implant - Dose 1 (low dose) (Experimental): Participants in Group 1 will receive a low dose of TimoD implant in the study eye on Day 1.
  Interventions: Drug: TimoD implant; Device: Injector system
- TimoD implant - Dose 2 (intermediate dose) (Experimental): Participants in Group 2 will receive an intermediate dose of TimoD implant in the study eye on Day 1 if all participants in Group 1 have completed a 4-week treatment period with the lowest dose of TimoD implant and providing there are no safety issues in Group 1.
  Interventions: Drug: TimoD implant; Device: Injector system
- TimoD implant - Dose 3 (high dose) (Experimental): Participants in Group 3 will receive a high dose of TimoD implant in the study eye on Day 1 if all participants in Group 2 have completed a 4-week treatment period with the intermediate dose, providing there are no safety issues in Group 2.
  Interventions: Drug: TimoD implant; Device: Injector system

INTERVENTIONS:
Drug: TimoD implant — Consists of 1 TimoD implant administration in the study eye.
  Other Names: intraocular implant releasing timolol; investigational drug
Device: Injector system — This is a CE-marked injector intended for intraocular lens (IOL) delivery. In this study, the injector is used as an"intraocular implant injection system" outside of its scope of intended use.
  Other Names: ACCUJECT™ 2.2.-BL; Investigational device

SUMMARY:
The goal of this clinical trial is to test a new method to deliver an approved medicine called Timolol in the eye of participants with glaucoma or ocular hypertension and requiring cataract surgery.

The main questions it aims to answer are how safe are three different doses of the investigational drug is and how the body tolerates it.

The study will also check:

* how safely the implant is placed in and removed from the eye and how the body responds to the procedure,
* if and the amount of Timolol released in the bloodstream,
* if there is any positive effect on the pressure inside the eye.

DETAILED DESCRIPTION:
Timolol will be delivered through an investigational drug called 'TimoD implant'.

This implant is placed inside one eye, the study eye, with the help of an instrument (investigational device) called an injector system. This procedure will be performed in conjunction with the cataract surgery.

Three dose ranges of TimoD implant will be tested (low, intermediate, and high) in 3 groups of 6 participants.Participants will receive only one dose. The Timolol will be released slowly through the implant for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent.
* In good general and mental health without ongoing clinically significant abnormalities in medical history.
* Open-angle glaucoma or ocular hypertension and age-related cataract eligible for intra-capsular IOL placement.
* successful, uncomplicated cataract surgery

Exclusion Criteria:

* Subjects with a history of hypersensitivity or contraindications to β- blockers.
* Participants using any systemic or topical drug known to interfere with visual performance, pupil dilation, or iris structure
* Significant risks caused by washout of ocular hypotensive medications.
* Clinically significant ocular pathology other than OHT, glaucoma and cataract

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number (%) of participants experiencing adverse events | From Screening (up to Day -41) to end of study (Month 13)
Number (%) of participants experiencing adverse events of special interest (AESI) | From Screening (up to Day -41) to end of study (Month 13)

CONTACTS AND LOCATIONS:
Locations (1):
- Panama Eye Center, Panama City, Panama